CLINICAL TRIAL: NCT00163254
Title: Balloonangioplasty or Stents With ReoPro for Prevention of Subacute Reocclusion in Arteries Below the Knee
Brief Title: Below Study - Balloonangioplasty or Stents With ReoPro for Prevention of Subacute Reocclusion in Arteries Below the Knee
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: btk-1; D 30.08290
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Patients Above 18 Years
Keywords: Chronic limb ischemia; Intervention; Restenosis; Patients above 18 years
MeSH Terms: interventions — Abciximab; Drug-Eluting Stents

INTERVENTIONS:
Drug: abciximab
Device: stent and drug eluting stent

SUMMARY:
The Below-Study is a randomized, prospective mono-centre trial on the efficacy and safety the adjunctive use of a GP IIb/IIIa antagonist for prevention of early reocclusion in arterial below-the knee interventions.

DETAILED DESCRIPTION:
PTA below the knee is limited due to subacute reocclusions and uncertain long-term results. This study is designed as a feasibility trial, which compares the two new treatment modalities: drug eluting stents and GP IIb/IIIa blockade.

Patients with current ulcers (Rutherford 5, or 6) are randomly assigned to one of the treatment groups: [1] ReoPro + Sirolimus coated stent, [2] ReoPro + bare Stent, [3] ReoPro + PTA, [4] PTA without ReoPro. Angiographic control will be at 2 and 6 months with block wise randomisation to the treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of peripheral artery disease with below the knee artery occlusion, or stenosis which mandates PTA or stent administration as first treatment modality. The history of peripheral artery occlusion has to at least 6 weeks, and the target vessel occlusion has to be no longer than 5 centimeters in length (corresponding to a maximum of 2 stents per treated lesion). The number of treated lesions per vessel in this study is limited to three. Only the major lesion will be allocated to one of the study groups, the other lesions will be treated by conventional PTA. A documentation of distal outflow (no occlusion until 3 cm above the upper joint ankle) is mandatory
* Severe stage of PAD with ulceration(s) corresponding to Rutherford stage 5 or 6.

Exclusion Criteria:

* Acute limb ischemia
* Subacute ischemia with requires thrombolysis as first treatment modality
* Active bleeding or known bleeding diathesis
* Known severe hepatic or renal disorder (liver cirrhosis, stage B, C or serum creatinine > 2.5 mg%)
* Hyperthyreosis
* Diabetes mellitus treated with metformin
* Known heparin induced thrombocytopenia (HIT, type 2)
* Major surgery, eye surgery or trauma within past 6 weeks
* History of stroke within the previous 2 years, or any stroke with a residual neurological deficit, or other CNS abnormality (e.g., intracranial neoplasm, arteriovenous malformation, or aneurysm), or history of aneurysm repair
* Gastrointestinal or genitourinary bleeding of clinical significance within the previous 6 weeks
* Puncture of a non compressible vessel within past 24 hours
* Administration of oral anticoagulants within the previous 7 days unless prothrombin time is < 1.2 times control (or international normalized ratio [INR] <1.4), or ongoing treatment with oral anticoagulants
* History of bleeding diathesis of platelet count < 100,000/mm3
* Known ReoPro-induced thrombocytopenia
* Arteriovenous malformations or aneurysms
* Severe uncontrolled hypertension (treated sys. BP > 200 mm Hg, diast. BP > 100 mm Hg)
* Known autoimmune disorders
* Patient with vasculitis
* Patient with aspirin intolerance
* Contraindication or known allergic reactions to rapamycin, abciximab or murine proteins
* Co-existent condition associated with a limited life expectancy (e.g., advanced cancer, end-stage congestive heart failure)
* Women of child-bearing potential with a positive pregnancy test
* Patient in prison or any vulnerable patient (soldier,…) as defined in the declaration of Helsinki

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Study Completion 2006-11

PRIMARY OUTCOMES:
The primary study objective is to demonstrate the superiority of an adjunctive administration of abciximab and drug eluting stents on the rate of subacute reocclusions at day 60 ± 10.

SECONDARY OUTCOMES:
The binary restenosis rate (restenosis > 50%) at 6 months
The rate of mortality, amputation (including toes), repeat target vessel intervention, and healing of ulcers 2 and 6 months from randomization.
Quality of life assessment 2 and at 6 months compared to baseline
Change in ankle brachial index (ABI) after the intervention, at 2 and at 6 months.
Change in Rutherford stages at 2 and at 6 months compared to baseline.
Hospital days for index hospitalization
Hospital days for repeat revascularization and amputation at 2 and 6 months
Safety analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Tübingen, Germany